CLINICAL TRIAL: NCT03722394
Title: Pain Neuroscience Education for Acute and Sub-Acute Low Back Pain: An Exploratory Case Series
Brief Title: Pain Neuroscience Education for Acute and Sub-Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Project Coordinator, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1202-4022
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain; Pain, Chronic; Pain, Back
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: Observational cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Neuroscience Education (Experimental): Subjects received a 15-minute verbal, one-on-one Pain Neuroscience Education (PNE) session
  Interventions: Behavioral: Pain Neuroscience Education

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — 15 minute verbal one-on-one education session

SUMMARY:
To determine if Pain Neuroscience Education (PNE) would result in positive clinical changes in patients presenting with acute or sub-acute low back pain (LBP).

DETAILED DESCRIPTION:
Background: Pain neuroscience education (PNE) has shown efficacy in treating chronic pain. Clinicians may believe PNE is not suitable for acute and sub-acute pain. Subgroupings of low back pain (LBP) imply some patients with LBP may respond favorably to PNE.

Objective: To determine if PNE would result in positive clinical changes in patients presenting with acute or sub-acute LBP.

Methods: Eighty consecutive patients with LBP < 3 months were enrolled in the study. Patients completed a demographics questionnaire, leg and LBP rating (Numeric Pain Rating Scale - NPRS), disability (Oswestry Disability Index), fear-avoidance (Fear-Avoidance Beliefs Questionnaire), pain catastrophization (Pain Catastrophization Scale), central sensitization (Central Sensitization Inventory), pain knowledge (Revised Neurophysiology of Pain Questionnaire), risk assessment (Keele STarT Back Screening Tool), active trunk flexion and straight leg raise (SLR). Patients received a 15-minute verbal, one-on-one PNE session, followed by repeat measurement of LBP and leg pain (NPRS), trunk flexion and SLR.

ELIGIBILITY:
Inclusion Criteria:

* a complaint of LBP with or without leg pain less than 3 months, and
* a willingness to participate

Exclusion Criteria:

* a) were under age 18 (minor);
* b) had undergone lumbar surgery;
* c) could not read or understand the English language;
* d) presented with any cognitive deficits rendering them unsuitable for PNE (i.e., stroke, traumatic brain injury, etc.),
* e) declined to participate or
* f) presented with a medical etiology (red flag) associated with their LBP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
NPRS - LBP | Immediate change from baseline after assigned intervention
  Numeric Pain Rating Scale for Low Back Pain (Range 0 = no pain to 11 = maximum pain)
NPRS - Leg pain | Immediate change from baseline after assigned intervention
  Numeric Pain Rating Scale for leg pain (Range 0 = no pain to 11 = maximum pain)

SECONDARY OUTCOMES:
Active trunk flexion | Immediate change from baseline in centimeters after assigned intervention
  Active trunk flexion measured in centimeters from fingertips to floor
Passive Straight Leg Raise | Immediate change from baseline in angular degrees after assigned intervention
  Range of hip flexion angle during passive straight leg raise test measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, PhD, Principal Investigator — St. Ambrose University
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No